CLINICAL TRIAL: NCT06371196
Title: Clinical Study on the Treatment of Elevated Total Bilirubin in Primary Biliary Cholangitis With Baobao Dan Capsule
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mei Han (Other)
Responsible Party: Sponsor-Investigator, Mei Han, Principal Investigator, Beijing University of Chinese Medicine
Organization: Beijing University of Chinese Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBD-PBC 2024-03
Record Dates: First submitted 2024-03-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Babaodan Capsule (Experimental): Babaodan Capsule (State Drug License: Z10940006) is manufactured by Xiamen Traditional Chinese Medicine Factory Co., Ltd; Packing specification: 0.3g/capsule, 6 capsules/board×2 boards/carton; Ingredients are in vitro cultivated cowhide, snake gallbladder, antelope horn, pearl, panax ginseng, artificial musk and so on.
  Interventions: Drug: Babaodan Capsule

INTERVENTIONS:
Drug: Babaodan Capsule — Babao Dan Capsule (State Drug License: Z10940006) is produced by Xiamen Traditional Chinese Medicine Factory Co., Ltd; Packing specification: 0.3g/capsule, 6 capsules/board×2 boards/small box; Ingredients are in vitro cultivated cowhide, snake gallbladder, antelope horn, pearl, panax ginseng, artificial musk, and so on. Intervention measures are really the original UDCA treatment program based on the addition of eight treasure Dan capsule, 2 capsules / times, tid, oral. Course of treatment: 3 months (based on 30 days/month).

SUMMARY:
1. Explore the effect of Babaodan Capsule on the serum total bilirubin level of primary biliary cholangitis patients with elevated total serum bilirubin;
2. To observe the positive intervention effect of Babaodan Capsule on the clinical symptoms of primary biliary cholangitis patients with elevated total bilirubin.

DETAILED DESCRIPTION:
1. Primary objective: to investigate the effect of Baobao Dan capsule on serum total bilirubin levels in patients with primary biliary cholangitis with elevated total serum bilirubin.
2. Secondary objective: to observe the effects of Babaodan Capsule on the following aspects in patients with primary biliary cholangitis with elevated total bilirubin:

(1) Other indicators of liver function: ALP, GGT, AST, ALT, TBA, TBil, DBil, IBil; (2) Itching and fatigue symptom scores; (3) Biochemical response rate; (4) Histologic changes; (5) Changes in immunologic indices (serum IgM, IgG, IgA, autoantibodies AMA/AMA-M2 and anti-gp210 antibody, anti-sp100 antibody); (6) Adverse events and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1. meets the diagnostic criteria for primary biliary cholangitis (PBC) in the Diagnostic and Therapeutic Guidelines for Primary Biliary Cholangitis (2021), i.e., meets at least 2 out of the following 3 criteria: (i) Biochemical evidence of cholestasis, i.e., elevated ALP and GGT, and imaging studies that exclude extrahepatic or intrahepatic biliary obstruction; (ii) Anti-mitochondrial antibody (AMA) or AMA-M2 positivity or, if AMA negative, PBC-specific antibody (anti-GP210 and/or anti-SP100) positivity; (iii) Histologic evidence suggestive of non-purulent destructive cholangitis and interlobular bile duct destruction.
* 2. Male or female, ≥ 18 years of age and < 75 years of age;
* 3. ursodeoxycholic acid capsule (Yusuf) 10 ~15 mg/d for ≥6 months prior to screening and after screening enrollment, the therapeutic dose was maintained unchanged for the duration of the trial;
* 4. ALP ≥ 1.67 x ULN;
* 5. liver function tests no less than 2 times in the last 3 months, and total bilirubin in liver function tests before enrollment and in the last 3 months are in accordance with the following: 1 × ULN < TBil ≤ 5 × ULN;
* 6. Understand the content of the study, be willing to comply with the study protocol, and voluntarily sign the written informed consent.

Exclusion Criteria.

* 1. Combination of or history of other liver diseases, including: (1) hepatitis C virus (HCV) infection; (2) hepatitis B virus (HBV) infection; (3) primary sclerosing cholangitis (PSC); (4) alcoholic liver disease; (5) autoimmune hepatitis (AIH) or overlapping autoimmune liver disease; (6) nonalcoholic steatohepatitis (NASH); (7) drug-induced liver injury; (8) extrahepatic biliary obstruction; (9) Gilbert's syndrome; (10) suspected or diagnosed primary liver cancer; (11) suspected or confirmed primary liver cancer; and (12) extrahepatic biliary obstruction; ⑨ Gilbert's syndrome; ⑩ suspected or confirmed primary liver cancer;
* 2. Presence of clinical complications of PBC, including but not limited to: (i) history of liver transplantation, pending liver transplantation, or current Model for End-Stage Liver Disease (MELD) score ≥ 15; (ii) portal hypertension with complications, including gastric or large esophageal varices, refractory or diuretic-resistant ascites, history of variceal hemorrhage, history of variceal treatment such as use of β-blockers, endoscopic tissue adhesive injections or ligatures, transjugular portacaval shunts, or hepatic encephalopathy; (iii) cirrhosis with Complications, including spontaneous bacterial peritonitis, hepatocellular carcinoma; 4. Hepatorenal syndrome (type I or II) or screening serum creatinine (Cr) ≥ 1.5 x ULN and serum creatinine clearance < 60 mL/min;
* 3. Hepatic function Child-Pugh classification grade B/C;
* 4. ALT ≥ 5 × ULN and/or AST ≥ 5 × ULN;
* 5. ALP > 10 × ULN;
* 6. patients with pruritus with severe itching or requiring systemic medication (e.g., bile acid sequestrants or rifampicin, etc.) within 2 months prior to enrollment
* 7. use of the following medications within 3 months prior to enrollment: azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, hexacosanol, dicyclomine, simethicone, ximethicone; fenofibrate or other fibrates; budesonide and other systemic corticosteroids; and hepatotoxic medications (including alpha-methyldopa, valproate, isoniazid, furosemide, etc.);
* 8. use of the following medications within 12 months prior to enrollment and throughout the trial: antibodies or immunotherapies against interleukins or other cytokines or chemokines;
* 9. having or having had a previous cardiac arrhythmia requiring clinical intervention that may affect survival during the trial; or pre-treatment QT prolongation or QTc intervals ≥470ms in men and ≥480ms in women
* 10. pregnant, planning pregnancy, breastfeeding women, women of childbearing potential who do not wish to use effective contraception (≥1 effective method of contraception e.g., condom, hormonal contraceptive pill, intrauterine device), or male subjects who do not wish to use contraception during the trial period and up to 30 days after the last dose of study medication
* 11. patients with co-infections of infectious diseases such as HIV, syphilis, and neo-coronavirus;
* 12. the presence of any other disease or condition that interferes with the absorption, distribution, metabolism, or excretion of the drug (e.g., patients with inflammatory bowel disease or those who have undergone gastric bypass surgery);
* 13. any other disease that is not well controlled or for which the need for the drug is expected to change during the trial;
* 14. persons with a suspected or confirmed history of alcohol or drug abuse within 1 year prior to screening;
* 15. incapacitated or restricted persons;
* 16. subjects who have been enrolled in another study within 30 days prior to Screening
* 17. mentally unstable or incapacitated persons for whom the validity of informed consent or compliance with the trial is uncertain;
* 18. has had a malignant tumor in the last 5 years, with or without treatment and with or without evidence of local recurrence or metastasis;
* 19. the patient has taken Babao Dan capsule within 1 month prior to the trial;
* 20. who, in the opinion of the investigator, should not participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total bilirubin (TBil) reversion rate | 90 days
  Total bilirubin (TBil) reversion rate: cases with normal total bilirubin index after treatment/60 cases × 100%
Total bilirubin (TBil) efficacy rate | 90 days
  Total bilirubin (TBil) efficacy rate: total bilirubin index decreased by 1×ULN cases/60 cases×100% after treatment compared with before treatment.

SECONDARY OUTCOMES:
biological response rate | 90 days
  Biological response rate of UDCA combined with Baobao Dan capsule in the treatment of PBC: number of cases meeting the biochemical response standard criteria / 60 cases × 100%. Referring to the UDCA treatment of PBC proposed in the "Diagnostic and therapeutic standard of primary biliary cholangitis (2021)", ALP <1.67×ULN was used as the biochemical response standard.
ALT | 90 days
  The actual level of ALT was collected in the form of measured information.
AST | 90 days
  The actual level of AST was collected in the form of measured information.
ALP | 90 days
  The actual level of ALP was collected in the form of measured information.
TBA | 90 days
  The actual level of TBA was collected in the form of measured information.
DBil | baseline, 30 days, 60 days, 90 days
  The actual level of DBil was collected in the form of measured information.
IBil | 90 days
  The actual level of IBil was collected in the form of measured information.
5-D Pruritus Scale Score | 90 days
  Evaluation was performed according to the 5-D Pruritus Scale Score, which includes 5 aspects of site, duration, intensity, tendency, and impairment of life, with a total score of 5 to 25.
Fatigue section of the PBC-40 questionnaire | 90 days
  It was carried out using the entries of malaise in the Quality of Life Questionnaire for Patients with Primary Biliary Cholangitis (PBC-40), which consisted of 11 items that were categorized according to the degree of malaise as none, seldom, sometimes, often, and continually, with scores of 1, 2, 3, 4, and 5, respectively, and a total score of 11-55.
Immunological indicators - serum IgM | 90 days
  The actual level of serum IgM was collected in the form of measured information.
Immunological indicators - serum IgG | 90 days
  The actual level of serum IgG was collected in the form of measured information.
Immunological indicators - serum IgA | 90 days
  The actual level of serum IgA was collected in the form of measured information.
Immunological indicators - anti-gp210 antibody | 90 days
  The actual level of anti-gp210 antibody was collected in the form of measured information.
Immunological indicators - anti-sp100 antibody | 90 days
  The actual level of anti-sp100 antibody was collected in the form of measured information.
Immunological indicators - autoantibodies AMA/AMA-M2 | 90 days
  The actual level of autoantibodies AMA/AMA-M2 was collected in the form of measured information.
Histopathology of the liver - grading of inflammatory activity | Changes of 90 days from the baseline.
  Baseline liver puncture biopsy results were valid for 6 months prior to screening, allowing patients to refuse to provide a histologic sample of the liver. The grading of inflammatory activity was observed and changes in the frequency of each corresponding grade were analyzed.
Histopathology of the liver - staging of the degree of fibrosis | Changes of 90 days from the baseline.
  Baseline results of hepatic puncture biopsy were valid for 6 months prior to screening, allowing patients to refuse to provide a histologic sample of the liver. The staging of the degree of fibrosis was observed and changes in the frequency of each corresponding grade were analyzed.
12-lead electrocardiogram | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal 12-lead electrocardiogram.
Physical examination | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal physical examination which concludes general examination of the whole body, head examination, neck examination, chest examination, abdominal examination, etc.
Routine blood test | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal routine blood test which concludes RBC, Hb, HCT, MCV, MCHC, RDW, WBC, Neut, Lymph, Mono, Eos, Basso, PLT.
Renal Function Tests-BUN | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal BUN.
Renal Function Tests-UA | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal UA.
Renal Function Tests-Scr | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal Scr.
Urinalysis | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
Coagulation tests-PT | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal PT.
Coagulation tests-APTT | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal APTT.
Coagulation tests-TT | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal TT.
Coagulation tests-FIB | baseline, 30 days, 60 days, 90 days
  This is a safety outcome. The test operator needs to check the numbers of participants with abnormal FIB.
Urine beta-hCG pregnancy test | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
adverse event | baseline, 30 days, 60 days, 90 days, 100 days
  This is a safety outcome.
Body temperature | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
Heart rate | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
Number of breaths in 1 min | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
Blood pressure-Diastolic blood pressure(mmHg) | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.
Blood pressure-Systolic blood pressure(mmHg) | baseline, 30 days, 60 days, 90 days
  This is a safety outcome.

IPD SHARING:
Plan to Share IPD: No